CLINICAL TRIAL: NCT04181606
Title: Age Comparisons of Exercising Muscle O2 Supply in Healthy Adults: Effects of Esmolol Infusion
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: David N. Proctor, PhD (Other)
Responsible Party: Sponsor-Investigator, David N. Proctor, PhD, Professor of Kinesiology, Physiology, and Medicine, Penn State University
Organization: Penn State University (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 10736
Record Dates: First submitted 2019-11-26; First posted 2019-11-29 (Actual); Results first posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-04

CONDITIONS: Aging
Keywords: Esmolol hydrochloride; Exercise
MeSH Terms: conditions — Motor Activity | interventions — esmolol; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The participants, investigators, and data analysts (outcomes assessors) will be blinded to the treatment (drug) order. The care providers (research nurse and physician) will be aware of the treatment order for safety reasons i.e., they will be assessing heart rate, blood pressure and symptoms before, during, and after the infusion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Esmolol Infusion (Active Comparator): Drug: Esmolol Hydrochloride Dosage form: Intravenous Infusion Dosage/Frequency: 0.5 mg/(kg Fat Free Mass·min) for 3 min followed by a maintenance infusion of 0.25 mg/(kg Fat Free Mass·min) for remainder of trial, up to a maximum of 1 hour.
  Interventions: Drug: Esmolol infusion; Other: Pre exercise baseline; Other: Isometric handgrip exercise; Other: Semi-recumbent cycling
- Saline Infusion (Placebo Comparator): Saline infusion volume/rate matched to the calculated dose of esmolol.
  Interventions: Drug: Saline infusion; Other: Pre exercise baseline; Other: Isometric handgrip exercise; Other: Semi-recumbent cycling

INTERVENTIONS:
Drug: Esmolol infusion — The Esmolol loading dose will be 0.5 mg/kg fat free mass/min administered over the first 3 minutes, followed by a maintenance dose of 0.25 mg/kg fat free mass/min for the remainder of the protocol (maximum of 60 minutes).
  Other Names: Esmolol Hydrochloride
  Arms: Esmolol Infusion
Drug: Saline infusion — Saline will be rate/volume matched to the calculated esmolol dose.
  Other Names: Normal saline solution
  Arms: Saline Infusion
Other: Pre exercise baseline — Subject rests quietly while drug infusion begins (3 min loading dose followed by 10 min of maintenance dose) until heart rate and blood pressure stabilize.
Other: Isometric handgrip exercise — The subject will grip at 40% of their maximum and maintain that grip for 90 seconds. Once at rest and once during heavy intensity cycling.
Other: Semi-recumbent cycling — Subjects will pedal for 2-4 minutes at a very light intensity (20W), followed immediately by 5 minutes at a moderate intensity (at a workload intended to elicit 85% of the oxygen consumption observed at the lactate threshold), and 5 minutes of cycling at a heavy intensity (at a workload estimated to elicit oxygen consumption half way between those observed at the lactate threshold and respiratory compensation point). Subjects will then continue cycling at the heavy intensity for 90 seconds while performing isometric handgrip exercise.

SUMMARY:
This study will test the central hypothesis that postmenopausal women will demonstrate increased oxygen extraction in active leg muscle during leg cycling exercise while receiving an infusion of Esmolol, a fast-acting β1 selective antagonist, when compared to premenopausal women

DETAILED DESCRIPTION:
This study will test the central hypothesis that postmenopausal women will demonstrate increased oxygen extraction in active leg muscle during leg cycling exercise while receiving an infusion of Esmolol, a fast-acting β1 selective antagonist, when compared to premenopausal women. β1 selective antagonists (or "β1 blockers") are used to lower heart rate and improve O2 supply-to-demand balance in patients with coronary artery disease. By using esmolol to attenuate the central sympathetic response to exercise (increased heart rate and cardiac output) we can examine peripheral mechanisms of O2 delivery. The current project will evaluate how older postmenopausal women adjust active muscle O2 supply to an acute reduction in systemic O2 delivery during large muscle dynamic exercise when compared to younger premenopausal women.

ELIGIBILITY:
3.1 Inclusion Criteria

1. Capable of giving informed consent
2. Premenopausal women ages 18-35 years OR post-menopausal women ages 55-70 years
3. Satisfactory medical history and physical exam, as determined by a Clinical Research Center (CRC) clinician
4. Not currently taking medications affecting heart rate or contractility
5. Fluent in written and spoken English

3.2 Exclusion Criteria

Participants who will not be studied are those who:

1. Are less than 19 years of age or more than 70 years of age
2. Are pregnant or lactating
3. Are prisoners or institutionalized individuals or unable to consent
4. Diagnosed renal failure (Creatinine >2.0 mg/dl)
5. Diagnosed liver disease (ALT and aspartate aminotransferase {AST} 2 times normal)
6. Diagnosed Reynaud's disease
7. Have uncontrolled diabetes
8. Have uncontrolled hypertension
9. Have a left ventricular ejection fraction < 40%
10. Have a recent history of unstable angina or myocardial infarction (<6 months), unstable angina, or use of nitrate medications within past 2 weeks

10. Severe lung disease (i.e., on supplemental oxygen or frequently use rescue inhalers) 11. Diagnosed bleeding or clotting disorder or recent blood transfusion 12. Have asthma, history of thyroid issues or hyperkalemia 13. Known use of recreational drugs 14. Methylphenidate use

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-02-02 (Actual); Primary Completion 2023-04-25 (Actual); Study Completion 2023-04-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Noll Laboratory, University Park, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 37 Participants were screened for eligibility between February 2, 2022 and April 25, 2023 at the Clinical Research Center in University Park, Pennsylvania (PA). Of these, 30 were considered enrolled.
Pre-assignment Details: 30 participants were considered enrolled and 27 participants were randomized. The 3 participants who were not randomized dropped out of the study prior to the infusion visit.
Groups:
- Esmolol, Then Saline: Participants first received esmolol hydrochloride via intravenous infusion.
  Dosage/Frequency: 0.5 mg/(kg Fat Free Mass·min) for 3 min followed by a maintenance infusion of 0.25 mg/(kg Fat Free Mass·min) for remainder of trial, up to a maximum of 1 hour.
  After a washout period of 45 mins, they then received saline via intravenous infusion (volume/rate matched to the calculated dose of esmolol).
- Saline, Then Esmolol: Participants first received saline via intravenous infusion (volume/rate matched to the calculated dose of esmolol).
  After a washout period of 45 mins, they then received esmolol hydrochloride via intravenous infusion.
  Dosage/Frequency: 0.5 mg/(kg Fat Free Mass·min) for 3 min followed by a maintenance infusion of 0.25 mg/(kg Fat Free Mass·min) for remainder of trial, up to a maximum of 1 hour.
Period: First Intervention (up to 1 Hour)
Arm/Group | Esmolol, Then Saline | Saline, Then Esmolol
Started | 13 (6 younger, 7 older) | 14 (7 younger, 7 older)
Completed | 13 (6 younger, 7 older) | 14 (7 younger, 7 older)
Not Completed | 0 | 0
Period: Washout (45 Mins)
Arm/Group | Esmolol, Then Saline | Saline, Then Esmolol
Started | 13 (6 younger, 7 older) | 14 (7 younger, 7 older)
Completed | 13 (6 younger, 7 older) | 14 (7 younger, 7 older)
Not Completed | 0 | 0
Period: Second Intervention (up to 1 Hour)
Arm/Group | Esmolol, Then Saline | Saline, Then Esmolol
Started | 13 (6 younger, 7 older) | 14 (7 younger, 7 older)
Completed | 13 (6 younger, 7 older) | 14 (7 younger, 7 older)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Esmolol, Then Saline | Saline, Then Esmolol | Total
Number analyzed (Participants) | 13 | 14 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 24
  >=65 years | 1 | 2 | 3
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.0 (18.2) | 44.1 (18.2) | 44.6 (18.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 14 | 27
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 11 | 12 | 23
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 10 | 11 | 21
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 13 | 14 | 27

OUTCOME MEASURES:

1. Primary Outcome: Tissue Saturation Index (TSI) - Active Leg Muscle
Description: The primary outcome variable is the change in skeletal muscle oxygenation (∆TSI%) in the active leg muscle from baseline during recumbent cycling using near-infrared spectroscopy. TSI% represent the percentage of oxygenated hemoglobin relative to total hemoglobin in the tissue beneath the NIRS probe. Lower values represent a greater reduction in tissue oxygenation from baseline (greater oxygen extraction and/or reduced oxygen delivery).
  TSI% = oxy[heme] / total[heme] x 100
Time Frame: Last 60 seconds of Rest, Moderate exercise, and Heavy Exercise.
Population: 11 younger and 12 older at two different exercise intensities (Moderate and Heavy)
Measure: Mean (Standard Deviation); unit: % Total Labile Signal
Arm/Group | Esmolol Infusion | Saline Infusion
Number analyzed (Participants) | 23 | 24
% Total Labile Signal
  Younger - Moderate: number analyzed (Participants) | 11 | 12
  Younger - Moderate | -5.1 (3.2) | -3.1 (2.4)
  Younger - Heavy: number analyzed (Participants) | 11 | 12
  Younger - Heavy | -8.7 (3.5) | -6.3 (3.6)
  Older - Moderate: number analyzed (Participants) | 12 | 12
  Older - Moderate | -1.5 (0.9) | -0.5 (1.1)
  Older - Heavy: number analyzed (Participants) | 12 | 12
  Older - Heavy | -4.1 (2.7) | -2.8 (3.2)

2. Secondary Outcome: Tissue Saturation Index - Inactive Forearm Muscle
Description: The change in skeletal muscle oxygenation (∆TSI%) in the inactive forearm from baseline during recumbent cycling using near-infrared spectroscopy. TSI% represent the percentage of oxygenated hemoglobin relative to total hemoglobin in the tissue beneath the NIRS probe. Lower values represent a greater reduction in tissue oxygenation from baseline (greater oxygen extraction and/or reduced oxygen delivery).
  TSI% = oxy[heme] / total[heme] x 100
Time Frame: Last 60 seconds of Rest, Moderate exercise, and Heavy Exercise.
Population: 11 younger, 11 older
Measure: Mean (Standard Deviation); unit: % Total Labile Signal
Arm/Group | Esmolol Infusion | Saline Infusion
Number analyzed (Participants) | 22 | 22
% Total Labile Signal
  Younger - Moderate: number analyzed (Participants) | 11 | 11
  Younger - Moderate | -3.3 (2.5) | -1.3 (1.6)
  Younger - Heavy: number analyzed (Participants) | 11 | 11
  Younger - Heavy | -5.9 (4.5) | -2.3 (3.2)
  Older - Moderate: number analyzed (Participants) | 11 | 11
  Older - Moderate | -0.1 (2.3) | -0.5 (1.8)
  Older - Heavy: number analyzed (Participants) | 11 | 11
  Older - Heavy | -1.5 (2.8) | -0.4 (2.5)

3. Secondary Outcome: Systolic Blood Pressure
Description: Systolic Blood Pressure recorded via an automatic sphygmomanometer (SunTech Tango)
Time Frame: At rest and 3 minutes into moderate exercise and heavy exercise.
Population: 13 younger, 13 older
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Esmolol Infusion | Saline Infusion
Number analyzed (Participants) | 26 | 26
mmHg
  Younger - Rest: number analyzed (Participants) | 13 | 13
  Younger - Rest | 105 (9) | 104 (10)
  Younger - Moderate Intensity: number analyzed (Participants) | 13 | 13
  Younger - Moderate Intensity | 119 (9) | 137 (14)
  Younger - Heavy Intensity: number analyzed (Participants) | 13 | 13
  Younger - Heavy Intensity | 134 (8) | 156 (13)
  Older - Rest: number analyzed (Participants) | 13 | 13
  Older - Rest | 114 (16) | 116 (11)
  Older - Moderate Intensity: number analyzed (Participants) | 13 | 13
  Older - Moderate Intensity | 125 (12) | 145 (14)
  Old - Heavy Intensity: number analyzed (Participants) | 13 | 13
  Old - Heavy Intensity | 137 (14) | 173 (24)

4. Secondary Outcome: Heart Rate
Description: Heart rate recorded via EKG
Time Frame: Last 60 seconds of Rest, Moderate exercise, and Heavy Exercise.
Population: 13 Younger, 14 Older
Measure: Mean (Standard Deviation); unit: Beats/minute
Arm/Group | Esmolol Infusion | Saline Infusion
Number analyzed (Participants) | 27 | 27
Beats/minute
  Younger - Rest: number analyzed (Participants) | 13 | 13
  Younger - Rest | 64.5 (8.7) | 70.0 (11.1)
  Younger - Moderate Intensity: number analyzed (Participants) | 13 | 13
  Younger - Moderate Intensity | 106.3 (11.5) | 115.4 (16.4)
  Younger - Heavy Intensity: number analyzed (Participants) | 13 | 13
  Younger - Heavy Intensity | 123.1 (11.8) | 141.2 (18.0)
  Older - Rest: number analyzed (Participants) | 14 | 14
  Older - Rest | 60.5 (7.8) | 67.2 (11.7)
  Older - Moderate Intensity: number analyzed (Participants) | 14 | 14
  Older - Moderate Intensity | 89.9 (10.4) | 97.6 (13.0)
  Older - Heavy Intensity: number analyzed (Participants) | 14 | 14
  Older - Heavy Intensity | 105.5 (13.4) | 118.5 (20.6)

5. Secondary Outcome: Cardiac Output
Description: Cardiac Output recorded using bioimpedance cardiography
Time Frame: Last 60 seconds of Rest, Moderate exercise, and Heavy Exercise.
Population: 13 younger, 13 older
Measure: Mean (Standard Deviation); unit: Liters/minute
Arm/Group | Esmolol Infusion | Saline Infusion
Number analyzed (Participants) | 26 | 26
Liters/minute
  Younger - Rest: number analyzed (Participants) | 13 | 13
  Younger - Rest | 5.3 (0.9) | 5.9 (0.7)
  Younger - Moderate Intensity: number analyzed (Participants) | 13 | 13
  Younger - Moderate Intensity | 11.3 (2.2) | 12.6 (1.9)
  Younger - Heavy Intensity: number analyzed (Participants) | 13 | 13
  Younger - Heavy Intensity | 13.5 (2.0) | 15.9 (2.5)
  Older - Rest: number analyzed (Participants) | 13 | 13
  Older - Rest | 5.3 (0.8) | 5.8 (0.6)
  Older - Moderate Intensity: number analyzed (Participants) | 13 | 13
  Older - Moderate Intensity | 10.1 (1.6) | 11.0 (1.2)
  Older - Heavy Intensity: number analyzed (Participants) | 13 | 13
  Older - Heavy Intensity | 12.3 (1.7) | 14.1 (1.6)

6. Secondary Outcome: Diastolic Blood Pressure
Description: Diastolic Blood Pressure recorded via an automatic sphygmomanometer (SunTech Tango)
Time Frame: At rest and 3 minutes into moderate exercise and heavy exercise.
Population: 13 younger, 13 older
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Esmolol Infusion | Saline Infusion
Number analyzed (Participants) | 26 | 26
mmHg
  Younger - Rest: number analyzed (Participants) | 13 | 13
  Younger - Rest | 66 (8) | 63 (6)
  Younger - Moderate Intensity: number analyzed (Participants) | 13 | 13
  Younger - Moderate Intensity | 64 (8) | 59 (11)
  Younger - Heavy Intensity: number analyzed (Participants) | 13 | 13
  Younger - Heavy Intensity | 64 (8) | 62 (12)
  Older - Rest: number analyzed (Participants) | 13 | 13
  Older - Rest | 69 (9) | 69 (8)
  Older - Moderate Intensity: number analyzed (Participants) | 13 | 13
  Older - Moderate Intensity | 68 (6) | 68 (8)
  Old - Heavy Intensity: number analyzed (Participants) | 13 | 13
  Old - Heavy Intensity | 69 (6) | 68 (12)

7. Secondary Outcome: Mean Arterial Pressure
Description: Mean Arterial Pressure recorded via an automatic sphygmomanometer (SunTech Tango)
Time Frame: At rest and 3 minutes into moderate exercise and heavy exercise.
Population: 13 younger, 13 older
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Esmolol Infusion | Saline Infusion
Number analyzed (Participants) | 26 | 26
mmHg
  Younger - Rest: number analyzed (Participants) | 13 | 13
  Younger - Rest | 79 (7) | 77 (6)
  Younger - Moderate Intensity: number analyzed (Participants) | 13 | 13
  Younger - Moderate Intensity | 82 (7) | 85 (10)
  Younger - Heavy Intensity: number analyzed (Participants) | 13 | 13
  Younger - Heavy Intensity | 87 (7) | 93 (10)
  Older - Rest: number analyzed (Participants) | 13 | 13
  Older - Rest | 84 (11) | 85 (8)
  Older - Moderate Intensity: number analyzed (Participants) | 13 | 13
  Older - Moderate Intensity | 87 (7) | 94 (10)
  Old - Heavy Intensity: number analyzed (Participants) | 13 | 13
  Old - Heavy Intensity | 91 (8) | 103 (14)

8. Secondary Outcome: Stroke Volume
Description: Stroke Volume recorded using bioimpedance cardiography
Time Frame: Last 60 seconds of Rest, Moderate exercise, and Heavy Exercise.
Population: 13 younger, 13 older
Measure: Mean (Standard Deviation); unit: mL/beat
Arm/Group | Esmolol Infusion | Saline Infusion
Number analyzed (Participants) | 26 | 26
mL/beat
  Younger - Rest: number analyzed (Participants) | 13 | 13
  Younger - Rest | 84 (15) | 86 (13)
  Younger - Moderate Intensity: number analyzed (Participants) | 13 | 13
  Younger - Moderate Intensity | 107 (20) | 110 (17)
  Younger - Heavy Intensity: number analyzed (Participants) | 13 | 13
  Younger - Heavy Intensity | 110 (18) | 114 (19)
  Older - Rest: number analyzed (Participants) | 13 | 13
  Older - Rest | 88 (16) | 88 (17)
  Older - Moderate Intensity: number analyzed (Participants) | 13 | 13
  Older - Moderate Intensity | 113 (15) | 114 (14)
  Older - Heavy Intensity: number analyzed (Participants) | 13 | 13
  Older - Heavy Intensity | 117 (14) | 119 (16)

9. Secondary Outcome: Systemic Vascular Conductance
Description: Systemic Vascular Conductance recorded using bioimpedance cardiography
Time Frame: Last 60 seconds of Rest, Moderate exercise, and Heavy Exercise.
Population: 13 younger, 13 older
Measure: Mean (Standard Deviation); unit: mL/minute/mmHg
Arm/Group | Esmolol Infusion | Saline Infusion
Number analyzed (Participants) | 26 | 26
mL/minute/mmHg
  Younger - Rest: number analyzed (Participants) | 13 | 13
  Younger - Rest | 70 (13) | 82 (9)
  Younger - Moderate Intensity: number analyzed (Participants) | 13 | 13
  Younger - Moderate Intensity | 141 (27) | 154 (32)
  Younger - Heavy Intensity: number analyzed (Participants) | 13 | 13
  Younger - Heavy Intensity | 159 (28) | 179 (42)
  Older - Rest: number analyzed (Participants) | 13 | 13
  Older - Rest | 67 (8) | 72 (7)
  Older - Moderate Intensity: number analyzed (Participants) | 13 | 13
  Older - Moderate Intensity | 117 (14) | 118 (8)
  Older - Heavy Intensity: number analyzed (Participants) | 13 | 13
  Older - Heavy Intensity | 132 (15) | 136 (14)

10. Secondary Outcome: ∆HHb - Inactive Forearm
Description: Change in deoxygenated hemoglobin (∆HHb) in the inactive forearm muscle from baseline during recumbent cycling exercise using near-infrared spectroscopy (NIRS) relative to the Total Labile Signal.
  ∆HHb is an index of oxygen extraction obtained using NIRS. The total labile signal is defined as the difference between the highest observed HHb value during 5 minutes of limb occlusion at 250 mmHg and the lowest observed HHb value observed during reperfusion following removal of the occlusion.
  Greater ∆HHb values indicate greater oxygen extraction in the tissue under the NIRS probe.
Time Frame: Last 60 seconds of Moderate and Heavy Exercise
Population: 9 younger, 12 older
Measure: Mean (Standard Deviation); unit: % Total Labile Signal
Arm/Group | Esmolol Infusion | Saline Infusion
Number analyzed (Participants) | 21 | 21
% Total Labile Signal
  Younger - Moderate Exercise: number analyzed (Participants) | 9 | 9
  Younger - Moderate Exercise | 8.6 (5.7) | 5.0 (4.1)
  Younger - Heavy Exercise: number analyzed (Participants) | 9 | 9
  Younger - Heavy Exercise | 13.5 (10.0) | 5.9 (7.0)
  Older - Moderate Exercise: number analyzed (Participants) | 12 | 12
  Older - Moderate Exercise | 2.9 (6.5) | -3.4 (6.1)
  Older - Heavy Exercise: number analyzed (Participants) | 12 | 12
  Older - Heavy Exercise | 4.1 (9.1) | -2.6 (10.4)

ADVERSE EVENTS:
Time Frame: Participants were monitored for safety during the course of each study visit, up to 6 weeks. Duration of study visits varied, but never exceeded four hours in length. During the infusion visit, participants were monitored by a clinician from the start of infusion until blood pressure and heart rate returned to baseline levels following the end of the infusion. Infusion time never exceeded one hour.
Description: No adverse events.
Groups:
- Esmolol: Participants received esmolol hydrochloride via intravenous infusion.
  Dosage/Frequency: 0.5 mg/(kg Fat Free Mass·min) for 3 min followed by a maintenance infusion of 0.25 mg/(kg Fat Free Mass·min) for remainder of trial, up to a maximum of 1 hour.
- Saline: Participants received saline via intravenous infusion (volume/rate matched to the calculated dose of esmolol).
Arm/Group | Esmolol | Saline
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 0/27 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-10-17): https://cdn.clinicaltrials.gov/large-docs/06/NCT04181606/Prot_SAP_000.pdf
  • Informed Consent Form (2022-11-18): https://cdn.clinicaltrials.gov/large-docs/06/NCT04181606/ICF_001.pdf